CLINICAL TRIAL: NCT05322317
Title: Testing Critical Components for a Trial of Advance Care Planning in Primary Care for Dementia
Brief Title: Advance Care Planning (ACP) in Primary Care for Dementia
Acronym: ADVANCE-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Annette Totten, Associate Professor and Core Investigator of Medical Informatics and Clinical Epidemiology, School of Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00023109
Record Dates: First submitted 2022-03-10; First posted 2022-04-11 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Dementia; Advance Care Planning
Keywords: dementia; advance care planning; primary care; ECHO
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a prospective pilot study designed to achieve the objectives listed above. This project focuses on implementing ACP (which is an accepted best practice) and using ECHO (which is an evidence-based existing professional development model in healthcare). The research component involves data collection from clinicians and clinics in addition to what would be normally collected for as part of the training program and for quality improvement (QI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot participants (Other): Participants will participate in ADVANCE-PC training via ECHO and will receive practice facilitation support, if needed.
  To assess the feasibility of the ADVANCE-PC training and implementation support, research data will be collected from participating clinicians at three time points. Two data collection points will be pre and post ECHO program training questionnaires about attitudes, experience, and intentions related to ACP and dementia. The third will be an interview at the end of the follow-up period, focusing on barriers to and facilitators of ACP in the context of dementia and the impact of the training and implementation support. Feasibility and acceptability of this intervention will be evaluated using descriptive and qualitative analyses of these data.
  Interventions: Other: ADVANCE-PC training via ECHO

INTERVENTIONS:
Other: ADVANCE-PC training via ECHO — To assess the feasibility of using a technology-based platform to deliver the ADVANCE-PC program to multiple primary care clinics. This model will be based on the ECHO program, a tele-mentoring program which uses communications technology to provide facilitated education, case review, and peer-to-peer problem solving remotely. Our working hypothesis is that the use of ECHO will be efficient (allowing several clinicians and teams to be supported simultaneously while creating a community of practice), feasible (that clinicians will enroll and share experiences via mentoring, guidance, feedback, and didactic education), and have the potential to impact patients as clinicians perceptions shift to favor ACP, their skills increase, and they are able to integrate ACP for patients with dementia into their clinic.

SUMMARY:
ADVANCE-PC: Aligning Dementia & adVANce Care planning Education in Primary Care, is a communications and implementation support intervention that builds on existing ACP programs, understanding of dementia, and clinical expertise to provide training and technical assistance tailored to the needs of primary care clinicians and clinics that are often over-burdened and under-resourced. For this pilot, we will recruit six primary care clinics to test the ADVANCE-PC delivered using remote technology (ECHO). The pilot will include conducting one ECHO cycle and assessing the feasibility and acceptability of the program content and this mode of delivery (Aim 1) and testing pragmatic outcome assessment for the intervention (Aim 2).

DETAILED DESCRIPTION:
Aim 1: To assess the feasibility, acceptability, and content utility of the ECHO program among the clinicians in the participating primary care clinics. Data will be collected to assess successful program implementation and participant engagement. We will document outreach efforts, reporting why clinics decline to participate and as well as the initial motivations of those who agree. Data will be collected from participating clinicians: a pre-training questionnaire about their prior experience with ACP and dementia; feedback at the end of each session; and a longer questionnaire at the end of the training that measures intentions to engage in ACP, their understanding of dementia, their confidence in engaging patients and families in ACP, and what barriers they expect to encounter. Attendance will be documented, and ECHO sessions will be recorded so participation and trainee engagement can be assessed. At the end of the follow-up period, clinicians will participate in interviews focused on barriers to and facilitators of ACP in the context of dementia. Feasibility and acceptability of this intervention will be evaluated using descriptive and qualitative analyses of these data.

Aim 2: To pilot test the ascertainment of outcomes for the ADVANCE-PC program in the 3-month period when trained clinicians are attempting to conduct ACP routinely in their clinics. The primary outcome will be the proportion of patients with dementia and/or their care partners seen by participating clinicians who are engaged in ACP. To pilot test pragmatic assessment of this outcome, we will work with clinics to determine how the number of patients with dementia seen in a defined period (the denominator) and number who are engaged in ACP (the numerator) can be efficiently identified in by each clinic using their electronic health record (EHR). We will collect information on EHR functionality and current dementia and ACP documentation during Months 1-3 and integrate support for documentation and measurement into the training. Our secondary outcomes are clinician confidence, intentions, and behavior related to ACP. These will be evaluated during the ECHO program using questionnaires modeled after data collection activities routinely used by clinics for quality improvement and formally measured and analyzed using research questionnaires pre and post completion of the ECHO program and a semi structured interview at the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Clinic Level

The program will be offered to six primary care clinics. Each must meet the following criteria:

* Be a member in a practice-based research network (PBRN) within the Meta-network Learning and Research Center (Meta-LARC),
* Have a functional EHR,
* Have leadership that agrees to clinic participation, and
* Is willing to attempt to track and report the number of eligible patients (those with dementia seen in the clinic by program-trained clinicians) and the number of these patients and/or care partners that received ACP from these program-trained clinicians during a 5-month follow-up period.

Clinician/Staff Level

Within participating clinics, primary care clinicians and other staff must meet all the following inclusion criteria to participate in the training program and the research questionnaire/interview:

* Willing to participate in ECHO sessions,
* Willing to work on ACP implementation between sessions, and
* Be highly likely to have visits with at least 8 patients with dementia and/or their care partners in a 5-month follow-up period.

Adults of any age and pregnant people will be allowed to participate. Primary care clinicians and staff will all be over 18 years old and there is no maximum age limit for participation. It is possible that a primary care clinician or staff member who participates may be pregnant. This research does not inquire about pregnancy status and there is no added risk to the fetus in including a pregnant person in professional training.

Exclusion Criteria:

Anyone meeting one or more of the exclusion criteria listed here will be excluded. We will exclude:

* Children and adolescents, as the target population is primary care clinicians, patient care team members, and primary care clinic staff;
* Clinicians who do not provide primary care;
* Primary care clinicians who do not care for patients with dementia; and
* Primary care clinics that do not have sufficient clinicians (6 clinicians or team members) or sufficient patients (at least 8 patients each) with dementia to meet the pilot test targets.

There will be no systematic exclusion of participants based on age, gender or race, and/or ethnicity.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Percentage of enrolled participants who attend 80% of ECHO program sessions | 5 months after start of program
  number of participants who attended 80% of sessions/number of enrolled participants
Proportion of patients with dementia and/or their care partners seen by participating clinicians who are engaged in ACP. | 8 months after start of program
  Primary care clinics will identify: patients with dementia and/or their care partners who have visits with participating clinicians during the study period (denominator) and track the number of these people who are engaged in advance planning during the project period (numerator)

SECONDARY OUTCOMES:
Participating clinician satisfaction rating: questionnaire designed for this study | 8 months from start of ECHO program
  A score created by combining 3 items from our study questionnaire: willingness to recommend the program to others, rating of relevance to their practice, and satisfaction with program content.
Percentage of enrolled participants who plan to continue to engage patients with dementia in ACP | 8 months after start of program
  number of participants who respond Yes to an item on the project questionnaire that asks if they will continue with ACP.

CONTACTS AND LOCATIONS:
Overall Officials: Annette M Totten, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No